CLINICAL TRIAL: NCT06236776
Title: Arrhythmia Assessment in Structural Cardiac Interventions Using Wearable ECG Monitoring: AWARE Registry
Brief Title: AWARE Registry: Wearable ECG in Structural Heart Interventions
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2023-0031
Record Dates: First submitted 2023-11-10; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Atrial Septal Defect; Patent Foramen Ovale
MeSH Terms: conditions — Heart Septal Defects, Atrial; Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multi-center (Sinchon Severance hospital / Gangnam Severance hospital), prospective cohort observational study to patients who had undergone structural heart intervention including device closure for secundum type atrial septal defect or Patent foramen ovale. Transthoracic echocardiography will be performed before the procedure, immediately after, and at 6, 18, 30 months after the procedure. Wearable ECG monitoring (> 3 days) will be performed before the procedure or immediately after procedure. Demographic, laboratory, hemodynamic data during procedure, and non-invasive imaging dat are obtained.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 19 year-old
* Patients who scheduled to perform percutaneous device closure for atrial septal defect or patent foramen ovale
* Patients provided with the written, informed consent to participate in this study

Exclusion Criteria:

* Patients who had paroxysmal, persistent, or chronic AF
* Life expectancy < 12 months
* Subject who the investigator deems inappropriate to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who scheduled to perform percutaneous device closure for atrial septal defect or patent foramen ovale
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of atrial fibrillation | Immediate post-operative
  Occurrence of atrial fibrillation at Immediate post-operative, 18, and 30 month on wearable ECG monitoring
Occurrence of atrial fibrillation | 18 month
  Occurrence of atrial fibrillation at Immediate post-operative, 18, and 30 month on wearable ECG monitoring
Occurrence of atrial fibrillation | 30 month
  Occurrence of atrial fibrillation at Immediate post-operative, 18, and 30 month on wearable ECG monitoring

SECONDARY OUTCOMES:
All cause-death | Immediate post-operative, 18 month , 30 month
hospitalization for heart failure | Immediate post-operative, 18 month , 30 month
  hospitalization for heart failure: data from electronic medical record in Yonsei university health system
new atrial fibrillation | Immediate post-operative, 18 month , 30 month
new atrial tachycardia | Immediate post-operative, 18 month , 30 month
high burden of APC/PVC (>15%) | Immediate post-operative, 18 month , 30 month
  high burden of APC/PVC ( >15%): on wearable ECG monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Iksung Cho, Principal Investigator — Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University College of Medicine
Locations (1):
- Division of Cardiology, Yonsei University Health System, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No